CLINICAL TRIAL: NCT03045601
Title: Diagnostic Accuracy of Coronary Computed Tomographic Angiography Derived Fractional Flow Reserve Compared to Invasive Coronar Angiography With Fractional Flow Reserve
Brief Title: Diagnostic Accuracy of CT-FFR Compared to Invasive Coronar Angiography With Fractional Flow Reserve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2016/1609
Record Dates: First submitted 2017-01-26; First posted 2017-02-07 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2020-03

CONDITIONS: Coronary Disease
Keywords: Diagnostic Techniques, Cardiovascular; Coronary Angiography; Fractional Flow Reserve, Myocardial; Echocardiography, Stress
MeSH Terms: conditions — Coronary Disease | interventions — Echocardiography, Stress

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT-FFR (Experimental): Analyse With New CT-FFR Method
  Interventions: Diagnostic Test: CT-FFR
- Stress echocardiography (Active Comparator): Analyse With invasive FFR and stress echocardiography
  Interventions: Diagnostic Test: Stress echocardiography

INTERVENTIONS:
Diagnostic Test: CT-FFR — Invasive FFR and CCTA With CT-FFR
  Arms: CT-FFR
Diagnostic Test: Stress echocardiography — Stress echocardiography and invasive FFR
  Arms: Stress echocardiography

SUMMARY:
Invasive coronary angiography is currently considered gold standard in the assessment of coronary artery disease although the method has limitations. Most importantly invasive angiography only depicts coronary anatomy without determining its physiological significance i.e the likelihood that the stenosis impedes oxygen delivery to the heart muscle. Fractional flow reserve (FFR) is a catheterization technique for assessing the physiological significance of a coronary artery lesion during invasive coronary angiography. Coronary computed tomographic angiography (CCTA) is a noninvasive imaging test that has become an alternative route to diagnosis for patients with suspected coronary artery disease. Computational fluid dynamics combined with anatomical models based on CCTA scans allows determination of coronary flow and pressure, and has emerged as a promising diagnostic modality called CT-FFR. In this Project New Mathematical algorithms are developed for computation of CT-FFR. The main objective of this study is to determine the diagnostic accuracy of CT-FFR values obtained by the new method compared with invasive coronary angiography with fractional flow reserve and state-of-the-art dobutamin stress echocardiography.

ELIGIBILITY:
Inclusion criteria

* Proven stenosis by CCTA that require further investigation with invasive coronary angiography i.e. patients with estimated stenosis ≥30- 50%.
* Informed consent

Exclusion Criteria:

* Patients with unstable coronary artery disease.
* Previously treated with PCI or coronary surgery.
* Severe renal impairment i.e. GFR <30ml / min
* Contrast allergy
* Contraindication to adenosine / nitroglycerin / beta-blocker
* BMI> 40
* Patients referred on the basis of technically unsuccessful CTA, motion artifact or similar

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
CT- FFR values by New Method as a dichotomous variable | 4 weeks
  Determining the diagnostic accuracy of CT-FFR values obtained by the new method compared with invasive coronary angiography with fractional flow reserve
Worsening regional wall motion abnormality | 4 weeks
  Determining the diagnostic accuracy of invasive FFR with comprehensive stress echocardiographic techniques

CONTACTS AND LOCATIONS:
Overall Officials: Petter Aadahl, MD, PhD, Study Director — Norwegian University of Science and Technology
Locations (1):
- St Olavs Hospital, Klinikk for hjertemedisin, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Braten AT, Fossan FE, Muller LO, Jorgensen A, Stensaeth KH, Hellevik LR, Wiseth R. Automated computed tomography-derived fractional flow reserve model for diagnosing haemodynamically significant coronary artery disease: a prospective validation study. Eur Heart J Imaging Methods Pract. 2024 Sep 30;2(3):qyae102. doi: 10.1093/ehjimp/qyae102. eCollection 2024 Jul. PMID 39450294
- [Derived] Tjellaug Braten A, Holte E, Wiseth R, Aakhus S. Dobutamine stress echocardiography after positive CCTA: diagnostic performance using fractional flow reserve and instantaneous wave-free ratio as reference standards. Open Heart. 2024 Sep 30;11(2):e002899. doi: 10.1136/openhrt-2024-002899. PMID 39349050